CLINICAL TRIAL: NCT07315386
Title: Catatonic Syndrome in Adult Patients at Basurto Hospital: A Descriptive Study of Incidence, Comorbidity, and Short-Term Outcomes
Status: Recruiting | Type: Observational
Sponsor: Beatriz Rodriguez Cabo (Other)
Responsible Party: Sponsor-Investigator, Beatriz Rodriguez Cabo, Professor, University of the Basque Country (UPV/EHU)
Organization: University of the Basque Country (UPV/EHU) (Other)
Other Study IDs: HUB271125
Record Dates: First submitted 2025-12-18; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Catatonia
MeSH Terms: conditions — Catatonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to assess the incidence, sociodemographic and clinical characteristics, treatment response, and short-term outcomes of adult patients with catatonic syndrome in the Bilbao area (Spain). Data will be collected from January 2024 to December 2025 from all patients aged 18 years or older diagnosed with catatonia of any etiology at Basurto University Hospital who provide informed consent to participate.

DETAILED DESCRIPTION:
Catatonic syndrome is a severe neuropsychiatric condition characterized by motor, behavioral, and speech abnormalities, frequently accompanied by autonomic and affective disturbances. Although historically conceptualized as a subtype of schizophrenia, current diagnostic classifications (DSM-5, ICD 11) recognize catatonia as a transdiagnostic syndrome that may occur in association with a wide range of psychiatric, neurological, metabolic, toxic, autoimmune and other medical conditions. Early recognition is clinically relevant, as catatonia is potentially reversible and timely treatment is associated with improved short-term outcomes.

Available epidemiological data indicate marked variability in the reported incidence and prevalence of catatonia across populations and clinical settings. Population-based studies from high-income countries (UK, USA) have reported incidence rates of approximately 4-5 catatonic episodes per 100,000 person-years. In contrast, studies conducted in acute psychiatric inpatient settings have described substantially higher prevalence rates, ranging from approximately 20% to over 40% of admitted patients.

In Spain, published data are limited to selected hospital-based subpopulations. Prevalence rates of approximately 8-9% have been reported in older adults assessed by liaison psychiatry services in general hospitals, while markedly higher rates have been described in specific psychiatric inpatient samples, including geriatric psychiatry wards (nearly 40%) and patients hospitalized for first-episode psychosis (approximately 20-25%). These findings highlight the influence of age, clinical setting, and underlying diagnosis on observed prevalence estimates.

To date, however, no studies have been conducted in Spain that systematically examine the incidence or prevalence of catatonic syndrome across an unselected adult hospital population, irrespective of underlying diagnoses or specific clinical subgroups. Consequently, the epidemiology and short-term clinical course of catatonia in a general hospital setting encompassing all medical and psychiatric services remain insufficiently characterized.

This prospective observational cohort study aims to address this gap by describing the incidence, sociodemographic and clinical characteristics, comorbidity profile, treatment response, and short-term outcomes of adult patients diagnosed with catatonic syndrome at Basurto University Hospital, a general university hospital providing secondary-level care to the Bilbao area (Spain). The study includes patients attended in any hospital service, including the emergency department and inpatient medical or psychiatric units.

All consecutive patients aged 18 years or older who are diagnosed with catatonia of any etiology during hospital care between 1 January 2024 and 31 December 2025 will be eligible for inclusion. The diagnosis of catatonia will be established according to DSM-5 criteria, requiring the presence of at least three characteristic catatonic signs identified through systematic clinical assessment. In addition, the Bush-Francis Catatonia Rating Scale (BFCRS) will be administered to support diagnostic assessment and severity quantification at presentation and during follow-up. Participants will be followed prospectively throughout their hospital stay, from diagnosis until medical discharge.

-

Hypotheses

Given the descriptive and observational nature of the study, the following hypotheses are formulated as expected patterns based on existing literature.

Primary hypothesis

-The incidence, sociodemographic characteristics, clinical presentation, comorbidity profile, treatment response, and short-term outcomes of catatonic syndrome observed in this study are expected to be broadly consistent with those reported in previous studies conducted in comparable healthcare settings.

Secondary hypotheses

* The incidence of catatonic syndrome in the adult hospital population is expected to fall within the range reported in population-based studies from high-income countries.
* The age distribution of catatonia is expected to show a bimodal pattern, with higher occurrence in early adulthood and later life.
* Hypokinetic presentations are expected to be more frequent than hyperkinetic or mixed forms in the hospital setting.
* Catatonic syndrome is expected to be associated with a heterogeneous range of underlying psychiatric and medical conditions, including affective and psychotic disorders as well as neurological and autoimmune conditions.
* Treatment with benzodiazepines is expected to be associated with a high rate of short-term clinical improvement.
* In the short term, catatonia is expected to be associated with an increased risk of medical complications related to immobility, without a marked increase in in-hospital mortality.

Study Variables

The following variables will be systematically collected and classified as primary and secondary variables.

Primary variable

-Annual incidence of catatonic syndrome, calculated as the number of new cases diagnosed at Basurto University Hospital per year divided by the reference population of the Bilbao catchment area, expressed as cases per 100,000 inhabitants per year.

Secondary variables

* Sociodemographic variables: age and sex.
* Catatonia-related variables: catatonia subtype (hypokinetic, hyperkinetic, or dyskinetic/mixed), BFCRS total score, and Global Clinical Impression scores at admission and discharge.
* Comorbidity variables: underlying psychiatric diagnoses and medical conditions, including neurological, autoimmune, metabolic, and toxic etiologies.
* Treatment-related variables: type of treatment administered (benzodiazepines, electroconvulsive therapy, or other pharmacological interventions) and response to benzodiazepine treatment (yes/no).
* Outcome variables: short-term clinical evolution categorized as complete recovery, incomplete recovery, lack of response, or death during hospitalization.
* Hospitalization-related variables: occurrence of medical complications during admission, length of hospital stay, and discharge destination.

Statistical Analysis

Statistical analysis will be primarily descriptive, in line with the observational design of the study. Incidence rates will be calculated annually and expressed per 100,000 inhabitants. Categorical variables will be summarized using frequencies and percentages, and quantitative variables will be described using appropriate measures of central tendency and dispersion. Missing data and losses will be documented and considered in the interpretation of results.

-

Ethical and Legal Considerations

The study will be conducted in accordance with the principles of the Declaration of Helsinki and with applicable national and European legislation governing biomedical research and the protection of personal data, including Regulation (EU) 2016/679 (General Data Protection Regulation), Spanish Organic Law 3/2018 on Personal Data Protection and Guarantee of Digital Rights, and Law 14/2007 on Biomedical Research.

The study protocol has been submitted for evaluation and approval by the corresponding Research Ethics Committee. Participation is voluntary, and refusal to participate or withdrawal from the study will not affect the medical care provided.

Clinical data will be collected from electronic medical records by authorized study personnel and subsequently pseudonymized prior to analysis. Identifiable data will be stored separately from the study database under restricted access and appropriate technical and organizational security measures.

Written informed consent will be obtained from participants or their legal representatives whenever clinically feasible. In cases of acute catatonia in which the patient lacks decision-making capacity at the time of diagnosis, informed consent will be sought once clinical recovery allows adequate understanding (deferred consent). In the event of in-hospital death before consent can be obtained, clinical data may be included in accordance with ethical committee guidance and applicable legal provisions, in order to minimize information bias.

The study does not involve any additional diagnostic procedures or therapeutic interventions beyond standard clinical care. No financial compensation is provided to participants, and no commercial funding is involved. Study results will be disseminated through scientific publications and presentations, ensuring full confidentiality of participant data.

ELIGIBILITY:
Inclusion Criteria

* Age ≥ 18 years at the time of hospital care.
* Diagnosis of catatonic syndrome established according to DSM-5 criteria.
* Patients attended at Basurto University Hospital in any clinical setting, including the Emergency Department or inpatient physical or psychiatric units.
* Diagnosis made during the study period, from 1 January 2024 to 31 December 2025.
* Catatonia of any etiology, including psychiatric, neurological, medical, metabolic, toxic, or autoimmune causes.
* Provision of informed consent by the patient or their legal representative, when clinically feasible; deferred consent accepted in cases of acute catatonia.

Exclusion Criteria

* Refusal to participate in the study by the patient or their legal representative.
* Withdrawal of informed consent at any point during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients aged 18 years or older who are attended at Basurto University Hospital, a general university hospital providing secondary-level care to the Bilbao area (Spain), and who are diagnosed with catatonic syndrome during routine hospital care. Eligible participants include patients evaluated in any clinical setting, including the Emergency Department and inpatient medical or psychiatric units. Catatonia is diagnosed according to DSM-5 criteria and supported by systematic clinical assessment and severity quantification using the Bush-Francis Catatonia Rating Scale. Patients with catatonia of any etiology are included, reflecting an unselected adult hospital population.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Annual incidence of catatonic syndrome | From 1 January 2024 to 31 December 2025
  Annual incidence of catatonic syndrome in the adult hospital catchment population, defined as the number of new cases of catatonia diagnosed according to DSM-5 criteria at Basurto University Hospital during the study period, divided by the reference population of the Bilbao area and expressed as cases per 100,000 inhabitants per year. Diagnosis will be supported by systematic clinical assessment and severity quantification using the Bush-Francis Catatonia Rating Scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Beatriz Rodriguez Cabo, Bilbao, Vizcaya, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cuevas-Esteban J, Serrat F, Iglesias-Gonzalez M, Motta N, Jimenez-Fernandez B, Vila-Badia R, Colomer-Salvans A, Serra-Arumi C, Cacho ND, Corbella-Sotil A, Butjosa A, Pardo M; PROFEP Group; Usall J. Catatonia in first-episode psychosis: prevalence and psychopathological association. BJPsych Open. 2025 Sep 23;11(5):e220. doi: 10.1192/bjo.2025.10834. PMID 40985102
- [Background] Cuevas-Esteban J, Iglesias-Gonzalez M, Rubio-Valera M, Serra-Mestres J, Serrano-Blanco A, Baladon L. Prevalence and characteristics of catatonia on admission to an acute geriatric psychiatry ward. Prog Neuropsychopharmacol Biol Psychiatry. 2017 Aug 1;78:27-33. doi: 10.1016/j.pnpbp.2017.05.013. Epub 2017 May 19. PMID 28533149
- [Background] Peralta V, Cuesta MJ. Motor features in psychotic disorders. II. Development of diagnostic criteria for catatonia. Schizophr Res. 2001 Mar 1;47(2-3):117-26. doi: 10.1016/s0920-9964(00)00035-9. PMID 11278128
- [Background] Smith JR, Lim S, Bindra S, Marler S, Rajah B, Williams ZJ, Baldwin I, Hossain N, Wilson JE, Fuchs DC, Luccarelli J. Longitudinal Symptom Burden and Pharmacologic Management of Catatonia in Autism With Intellectual Disability: An Observational Study. Autism Res. 2025 Feb;18(2):449-462. doi: 10.1002/aur.3315. Epub 2025 Jan 27. PMID 39866085
- [Background] Ramirez-Bermudez J, Medina-Gutierrez A, Gomez-Cianca H, Arias P, Perez-Gonzalez A, Lebrija-Reyes PA, Espinola-Nadurille M, Aguilar-Venegas LC, Ojeda-Lopez C, Restrepo-Martinez M, Bayliss L, Juarez-Jaramillo CA, Penaloza G, Rivas-Alonso V, Flores-Rivera J, Gomez-Amador JL, Rios C, Sachdev PS. Clinical Significance of Delirium With Catatonic Signs in Patients With Neurological Disorders. J Neuropsychiatry Clin Neurosci. 2022 Spring;34(2):132-140. doi: 10.1176/appi.neuropsych.18120364. Epub 2022 Jan 18. PMID 35040665
- [Background] Rogers JP, Pollak TA, Begum N, Griffin A, Carter B, Pritchard M, Broadbent M, Kolliakou A, Ke J, Stewart R, Patel R, Bomford A, Amad A, Zandi MS, Lewis G, Nicholson TR, David AS. Catatonia: demographic, clinical and laboratory associations. Psychol Med. 2023 Apr;53(6):2492-2502. doi: 10.1017/S0033291721004402. Epub 2021 Nov 2. PMID 35135642
- [Background] Luccarelli J, Kalinich M, Fricchione G, Smith F, Beach SR, Smith JR. Diagnostic and demographic factors of pediatric and adult catatonia hospitalizations: A 2016-2020 National Inpatient Sample Study. Acta Psychiatr Scand. 2024 Oct;150(4):234-244. doi: 10.1111/acps.13744. Epub 2024 Aug 8. PMID 39118275
- [Background] Funayama M, Koreki A, Takata T, Kurose S. Catatonia, bedridden status, choking, water intoxication, and suicide are involved in deaths of schizophrenia inpatients. Asian J Psychiatr. 2020 Jun;51:102054. doi: 10.1016/j.ajp.2020.102054. Epub 2020 Apr 8. No abstract available. PMID 32283511
- [Background] Funayama M, Takata T, Koreki A, Ogino S, Mimura M. Catatonic Stupor in Schizophrenic Disorders and Subsequent Medical Complications and Mortality. Psychosom Med. 2018 May;80(4):370-376. doi: 10.1097/PSY.0000000000000574. PMID 29521882
- [Background] Jaimes-Albornoz W, Serra-Mestres J. Prevalence and clinical correlations of catatonia in older adults referred to a liaison psychiatry service in a general hospital. Gen Hosp Psychiatry. 2013 Sep-Oct;35(5):512-6. doi: 10.1016/j.genhosppsych.2013.04.009. Epub 2013 May 15. PMID 23684045
- [Background] Pelzer AC, van der Heijden FM, den Boer E. Systematic review of catatonia treatment. Neuropsychiatr Dis Treat. 2018 Jan 17;14:317-326. doi: 10.2147/NDT.S147897. eCollection 2018. PMID 29398916
- [Background] Hirjak D, Fricchione G, Wolf RC, Northoff G. Lorazepam in catatonia - Past, present and future of a clinical success story. Schizophr Res. 2024 Jan;263:27-34. doi: 10.1016/j.schres.2023.02.015. Epub 2023 Feb 18. PMID 36805317
- [Background] Cuevas-Esteban J, Serrat F, Baladon L, Rabaneda-Lombarte N, Díez-Quevedo C, Iglesias- González M. Factor analysis and validation of the Bush Francis catatonia rating scale-Spain version. The European Journal of Psychiatry [Internet]. 2023 Oct 1 [cited 2023 Nov 20];37(4):100221. Available from: https://www.sciencedirect.com/science/article/pii/S0213616323000344
- [Background] Bush G, Fink M, Petrides G, Dowling F, Francis A. Catatonia. I. Rating scale and standardized examination. Acta Psychiatr Scand. 1996 Feb;93(2):129-36. doi: 10.1111/j.1600-0447.1996.tb09814.x. PMID 8686483
- [Background] Luccarelli J, Kalinich M, Rogers JP, Donovan AL, Smith FA, Beach SR, Smith JR. Emergency Department Presentations for Catatonia: A 2019-2021 National Emergency Department Sample Study. J Acad Consult Liaison Psychiatry. 2025 Sep-Oct;66(5):380-388. doi: 10.1016/j.jaclp.2025.08.006. Epub 2025 Aug 8. PMID 40784551
- [Background] Wilson JE, Niu K, Nicolson SE, Levine SZ, Heckers S. The diagnostic criteria and structure of catatonia. Schizophr Res. 2015 May;164(1-3):256-62. doi: 10.1016/j.schres.2014.12.036. Epub 2015 Jan 13. PMID 25595653
- [Background] Subramaniyam BA, Muliyala KP, Hari Hara S, Kumar Reddi VS. Prevalence of catatonic signs and symptoms in an acute psychiatric unit from a tertiary psychiatric center in India. Asian J Psychiatr. 2019 Aug;44:13-17. doi: 10.1016/j.ajp.2019.07.003. Epub 2019 Jul 5. PMID 31302436
- [Background] Idrees MB, Elmahdi AM, Alharbi HY, Adam I. Catatonia in an acute adult inpatient population in mental health units in Khartoum, Sudan: A cross-sectional study. World J Psychiatry. 2025 Mar 19;15(3):102529. doi: 10.5498/wjp.v15.i3.102529. eCollection 2025 Mar 19. PMID 40109984
- [Background] Luccarelli J, Smith JR, Kalinich M, Amad A, Rogers JP. The Population-Based Incidence and Prevalence of Catatonia. J Neuropsychiatry Clin Neurosci. 2025 Spring;37(2):160-162. doi: 10.1176/appi.neuropsych.20240072. Epub 2025 Jan 10. PMID 39789943
- [Background] Beach SR, Luccarelli J, Praschan N, Fusunyan M, Fricchione GL. Molecular and immunological origins of catatonia. Schizophr Res. 2024 Jan;263:169-177. doi: 10.1016/j.schres.2023.03.013. Epub 2023 Mar 23. PMID 36966063
- [Background] Walther S, Stegmayer K, Wilson JE, Heckers S. Structure and neural mechanisms of catatonia. Lancet Psychiatry. 2019 Jul;6(7):610-619. doi: 10.1016/S2215-0366(18)30474-7. Epub 2019 Jun 10. PMID 31196794
- [Background] Moyal M, Iftimovici A, Ghoul W, Plaze M, Chaumette B. Genetics of catatonia: a systematic review of case reports and a gene pathway analysis. Eur Psychiatry. 2025 May 22;68(1):e72. doi: 10.1192/j.eurpsy.2025.2458. PMID 40400398
- [Background] Dalmau J, Gleichman AJ, Hughes EG, Rossi JE, Peng X, Lai M, Dessain SK, Rosenfeld MR, Balice-Gordon R, Lynch DR. Anti-NMDA-receptor encephalitis: case series and analysis of the effects of antibodies. Lancet Neurol. 2008 Dec;7(12):1091-8. doi: 10.1016/S1474-4422(08)70224-2. Epub 2008 Oct 11. PMID 18851928
- [Background] Rogers JP, Pollak TA, Blackman G, David AS. Catatonia and the immune system: a review. Lancet Psychiatry. 2019 Jul;6(7):620-630. doi: 10.1016/S2215-0366(19)30190-7. Epub 2019 Jun 10. PMID 31196793
- [Background] Luccarelli J, Kalinich M, McCoy TH Jr, Fernandez-Robles C, Fricchione G, Smith F, Beach SR. The occurrence of catatonia diagnosis in acute care hospitals in the United States: A national inpatient sample analysis. Gen Hosp Psychiatry. 2022 Jul-Aug;77:141-146. doi: 10.1016/j.genhosppsych.2022.05.006. Epub 2022 May 24. PMID 35660679
- [Background] World Health, Organization (WHO). International Classification of Diseases, Eleventh Revision (ICD-11) [Internet]. 2019. Available from: https://icd.who.int/browse11
- [Background] American Psychiatric Association. Diagnostic and statistical manual of mental disorders (5th ed.) [Internet]. 5th edn. 2013 [cited 2025 June 22]. Available from: https://doi.org/10.1176/appi.books.9780890425596
- [Background] Emil Kraepelin. Psychiatrie: Ein Lehrbuch. 6th ed. 6th edn. Leipzig, Germany: J. A. Barth; 1899.
- [Background] Kahlbaum KL. Die Katatonie oder das Spannungsirresein: eine klinische Form psychischer Krankheit. Leipzig: Hirschwald; 1874.
- [Background] Rogers JP, Oldham MA, Fricchione G, Northoff G, Ellen Wilson J, Mann SC, Francis A, Wieck A, Elizabeth Wachtel L, Lewis G, Grover S, Hirjak D, Ahuja N, Zandi MS, Young AH, Fone K, Andrews S, Kessler D, Saifee T, Gee S, Baldwin DS, David AS. Evidence-based consensus guidelines for the management of catatonia: Recommendations from the British Association for Psychopharmacology. J Psychopharmacol. 2023 Apr;37(4):327-369. doi: 10.1177/02698811231158232. Epub 2023 Apr 11. PMID 37039129

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-11-13): https://cdn.clinicaltrials.gov/large-docs/86/NCT07315386/Prot_SAP_000.pdf